CLINICAL TRIAL: NCT00114023
Title: A Follow-up Study to Evaluate Actinic Keratosis Recurrence Rates One Year After Completion of the 1473-IMIQ Study
Brief Title: 1-Year Follow up to the 1473-IMIQ Study
Status: Completed | Type: Observational
Sponsor: Graceway Pharmaceuticals, LLC (Industry)
Other Study IDs: 1518-IMIQ
Record Dates: First submitted 2005-06-13; First posted 2005-06-14 (Estimated); Last update posted 2007-02-19 (Estimated); Status verified 2006-10

CONDITIONS: Keratosis
Keywords: AK; Imiquimod 5% cream; 3M Pharmaceuticals; Aldara; Actinic Keratosis
MeSH Terms: conditions — Keratosis; Keratosis, Actinic | interventions — Imiquimod

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Drug: Imiquimod 5% cream

SUMMARY:
This is a 1-year follow-up study to evaluate the long-term effects in subjects who completely cleared their actinic keratosis (AK) lesions in the 1473-IMIQ study. The 1473-IMIQ study evaluated the safety and effectiveness of imiquimod 5% cream compared to a placebo cream for the treatment of AK.

ELIGIBILITY:
Inclusion Criteria:

* Subject had to participate in the 1473-IMIQ Study AND have had 100% clearance of AK lesions

Exclusion Criteria:

* Did not use any topical preparations in the previous treatment area within 24-hours of the scheduled visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84
Dates: Start 2005-01

CONTACTS AND LOCATIONS:
Locations (1):
- Little Rock, Arkansas, United States